CLINICAL TRIAL: NCT05197907
Title: Influence of Manual Relaxation of the Diaphragm on the Tension of the Posterior Superficial Fascia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Roksana Wójcik, Director, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: N43/DBS/000115
Record Dates: First submitted 2021-12-27; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Diaphragm; Relaxation; Low Back Pain
Keywords: diaphragm; low back pain; deep tissue massage; diaphragm relaxation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diaphragm fascial release group. (Experimental): Ten minutes lasting fascial release techinques performed on diaphragm.
  Interventions: Procedure: Fascial release of diaphragm muscle.
- Classic massage group (Placebo Comparator): Ten minutes lasting classic massage performed on abdomen.
  Interventions: Procedure: Classic massage of the abdomen.

INTERVENTIONS:
Procedure: Fascial release of diaphragm muscle. — The intervention consists of deep tissue massage techniques and manual mobilization of the fascia performed within the diaphragm attachments in the area of the costal arches.
  Arms: Diaphragm fascial release group.
Procedure: Classic massage of the abdomen. — The intervention consists of selected classic massage techniques - mainly stroking (effleurage) - performed on the superficial layers of the abdominal region
  Arms: Classic massage group

SUMMARY:
The diaphragm performs many functions that are vital to the body as a whole. Some of them are not related only to ventilation. The diaphragm is part of the myofascial system in the human body. Therefore, the proper functioning of the diaphragm should be a significant element of physiotherapy, e.g. in patients reporting pain in the lumbosacral spine.

Considering the complex role of the diaphragm, it seems reasonable to investigate the influence of the mobilization of the diaphragm (aimed at reducing diaphragm tension) on the tension of the extensor muscles of the lumbar spine.

The assumption of this reserach is to investigate the correlation between the tension of the fascia in the area of the diaphragm to the tension of the muscles in the area of the lumbar spine. The fascial connections between the diaphragm and the muscles in the lumbar spine presented above suggest that the manual therapy performed within the diaphragm can effectively prevent the occurrence of pain, and might be a supportive measure in the treatment of pain in the spine.

The aim of the study is to investigate the corellation between the tension of the fascia within the diaphragm and the tension of the posterior superficial tape.

Research questions:

1. How does manual therapy in the area of the tendon attachments of the diaphragm affect the relaxation of the extensor muscles of the lumbar spine?
2. How can the therapy conducted only within the diaphragm, without interfering with the structures surrounding the spine, reduce the tension of the extensor muscles of the lumbar spine and, consequently, increase the range of its mobility in all planes?
3. How will the introduced therapy change the tidal volume of the lungs?

ELIGIBILITY:
Inclusion Criteria:

* age within 20-40 yrs,
* BMI within normal range (18.5-24.9)
* lack of abdominal obesity
* lack of chronic musculoskeletal conditions
* written, conscious consent

Exclusion Criteria:

* former abdominal surgery
* abdominal diseases (i.e. (np. kidney stones, ulcers, irritative bowel sindrome, etc.),
* pregnancy
* fever,
* tumors,
* blood hypertension,
* former surgery of respiratory system ,
* condition after surgical procedures in the area of the spine,
* the occurrence of pain in the spine in the 3 months preceding the research experiment,
* lack of conscious consent

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Assessemnt of change in muscle tension of selected muscles of lumbar region | Twice - before and immediately after the treatment procedure
  Assessment of muscle superficial electromyography will be performed with sEMG device NuTrac Alpha2E (NeuroTrac Ltd.) on the following muscles: multifidus, longissimus and iliocostalis.

SECONDARY OUTCOMES:
Assessment of change of range of motion of the lumbar spine. | Twice - before and immediately after the treatment procedure
  The range of motion of the lumbar spine will be performed with the digital inclinometer (Baseline)
Assessment of change in peak expiratory flow in one second (PEF1) | Twice - before and immediately after the treatment procedure
  The peak expiratory flow in one second will be performed with PF100 peakflometer (Microlife).

CONTACTS AND LOCATIONS:
Overall Officials: Bartosz Trybulec, PhD, Study Chair — Jagiellonian University
Locations (1):
- Jagiellonian University Medical College, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No